CLINICAL TRIAL: NCT01754090
Title: Digital Therapy: Evaluation of the Fully Automated Alcohol Intervention "Balance".
Brief Title: Testing the Efficacy of an Online Alcohol Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Håvar Brendryen, Research fellow. PhD., University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SERAF-BALANCE-1
Record Dates: First submitted 2012-12-17; First posted 2012-12-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Hazardous Drinking; Harmful Drinking
Keywords: alcohol; online intervention; hazardous drinking; harmful drinking; early intervention; behavior change intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Receives two interventions:
  1. Online screening and feedback.
  2. Online booklet.
  Interventions: Behavioral: Online screening and feedback; Behavioral: Online booklet.
- Extended follow-up (Experimental): Receives two interventions:
  1. Online screening and feedback.
  2. Online multi session follow-up.
  Interventions: Behavioral: Online screening and feedback; Behavioral: Online multi session follow-up

INTERVENTIONS:
Behavioral: Online screening and feedback — An online single session screening procedure including individualized normative feedback.
Behavioral: Online booklet. — An online booklet that covers general information about alcohol, its effect on the brain and the body, potential risks and harms of drinking, and an account of the threshold values of sensible drinking
  Arms: Usual care
Behavioral: Online multi session follow-up — An online multi session follow-up program (i.e., "Balance"). The central concept of Balance is to support continued self-regulation throughout the behavior change process. There are four key aspects of the program, the first is focus on goal setting and tracking of alcohol consumption on a day-to-day basis. The second on relapse prevention - for example, when clients report drinking more than their target, they receive individualized content aimed at preventing a full blown relapse. The third is emotion regulation, where content and assignments from positive psychology and from cognitive behavioral therapy are used. Finally, intervention covers alcohol education (i.e. the same topics as in the booklet provided to the control group).
  Arms: Extended follow-up

SUMMARY:
The purpose of this study is to test whether an online multi session alcohol intervention improves treatment effect compared to single session screening with feedback only.

All participants in the trial received a single session screening procedure including individualized normative feedback (usual care). Additionally, half of the participants received a simple online booklet about the effects of alcohol. The other half received an online multi session follow up program.

DETAILED DESCRIPTION:
Aims: Test whether a multi session alcohol intervention improves treatment effect (i.e., reduced consumption of alcohol) compared to single session screening with feedback.

Design: Randomized controlled trial (RCT). Subjects in both conditions receives a single session screening procedure including individualized normative feedback. The control group receives an online booklet about the effects of alcohol. The treatment group receives the multi session follow up program "Balance" .

Setting: Online study in Norway. Participants: At-risk drinkers is recruited through internet advertisements and randomly assigned to one of two conditions.

ELIGIBILITY:
Inclusion Criteria:

* hazardous or harmful drinking (i.e., a FAST-score of 3 or more)

Exclusion Criteria:

* underage (<18)
* not provided a valid e-mail address
* not provided a valid (Norwegian) mobile phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
number of standard alcohol units consumed during the previous seven days | measures six months after baseline (enrollment)
  Subjects are asked to indicate (through online questionnaires) how many standard alcohol units they consumed on each of the previous seven days, on a scale from zero to ten. Then a sum-score for weekly consumption is calculated, ranging from zero to 70.

SECONDARY OUTCOMES:
Sick leave during last week | Assessed at six months post baseline
  Sick leave was assessed with a "yes" or "no" response for each of the past seven days, and then accumulated, resulting in a score of zero to seven. Participants were instructed to report any sick leave regardless of reason.
Negative consequences of alcohol consumption | Assessed at six months post baseline
  Perceived negative consequences of own alcohol consumption, during the seven previous days, was assessed by a 13 item index, resulting in a sum score with a theoretical range from zero to 13. The items comprised: headache, nausea, anxiety, worn out, depressed, breaking a plan, breaking a date, sick leave, memory problems, bad conscience, conflict, destroyed something and injuries.
Change in alcohol consumption | Six months post baseline
  The change score for weekly consumption, from baseline to six months, is calculated based on the seven day consecutive measure (primary outcome).
Number of days with alcohol consumption | Six months post baseline
  Based on the seven day consecutive measure (primary outcome), the number of days with alcohol consumption is calculated.
Number of alcohol binges | Six months post baseline
  Based on the seven day consecutive measure (primary outcome), the number of days with a binge drinking episode is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Håvar Brendryen, PhD, Principal Investigator — Norwegian Centre for Addiction Research, University of Oslo
Locations (1):
- Norwegian Centre for Addiction Research, University of Oslo, Oslo, Norway

REFERENCES:
- [Background] Brendryen H, Lund IO, Johansen AB, Riksheim M, Nesvag S, Duckert F. Balance--a pragmatic randomized controlled trial of an online intensive self-help alcohol intervention. Addiction. 2014 Feb;109(2):218-26. doi: 10.1111/add.12383. Epub 2013 Nov 21. PMID 24134709